CLINICAL TRIAL: NCT02219568
Title: Efficacy of Wireless Capsule Endoscopy and CT Enterography in Obscure Gastrointestinal Bleeding : Prospective Blinded Comparative Study
Brief Title: Efficacy of Wireless Capsule Endoscopy and CT Enterography in Obscure Gastrointestinal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Julajak Limsrivilai, Instructor in Internal medicine, Gastroenterlogy Division, Siriraj Hospital, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si624/2013
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Gastrointestinal Bleeding
Keywords: obscure gastrointestinal bleeding, CT enterography
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Capsule Endoscopy

ARMS (1):
- obscure gastrointestinal bleeding (Experimental): Those patients who developed obscure gastrointestinal bleeding either overt or occult bleeding who will then undergo video capsule endoscopy and CT enterography.
  Interventions: Procedure: CT enterography; Device: video capsule endoscopy

INTERVENTIONS:
Procedure: CT enterography — CT enterography is performed using 64-channel multi-detector row CT scanners (Siemens Sensation 64, Siemens Medical solution, Forchiem, Germany). Prior to the scan, 1500 cc of a neutral oral-enteric contrast material, polyethylene glycol (NIFLEC) is taken by the patient. During the scan, 2cc/kg of intravenous contrast (iohexol, Ominipaque Amersham GE-Health care, Princeton, NJ) is injected at the velocity 5 cc/sec.
Device: video capsule endoscopy — Video capsule endoscopy is performed using PillCam SB (Given Imaging, Yokneam, Israel). Polyethylene glycol (NIFLEC) is used for bowel preparation.

SUMMARY:
The purpose of this study is to compare the efficacy between video capsule endoscopy and CT enterography in diagnosis of obscure gastrointestinal bleeding.

DETAILED DESCRIPTION:
All adult patients with obscure gastrointestinal bleeding will undergo both video capsule endoscopy and CT enterography. The interval between two tests will be less than 1 month. The capsule reading gastroenterologist and the CT reading radiologist are blinded to each others' results.

ELIGIBILITY:
Inclusion Criteria:

* patients who present with passing melena or hematochezia or have iron deficiency anemia
* no lesion found on both esophagogastroduodenoscopy and colonoscopy
* age at least 18 years

Exclusion Criteria:

* allergy to iodinated intravenous contrast
* chronic kidney disease stage at least 3 patients who do not on regular dialysis
* suspected small bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
number of significant gastrointestinal lesions detected | up to 1 month
  Significant gastrointestinal lesions are ulcers, mucosal inflammation, angiodysplasia, and mass.

CONTACTS AND LOCATIONS:
Overall Officials: Julajak Limsrivilai, M.D., Principal Investigator — Mahidol University
Locations (1):
- Gastroenterology division, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand